CLINICAL TRIAL: NCT00338052
Title: Open-Label Study of Cycle Control With Extended Administration of Norethindrone Acetate 1 mg / Ethinyl Estradiol 20 Mcg Oral Tablets
Brief Title: Study of Bleeding With Extended Administration of an Oral Contraceptive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Herman Ellman, MD, Warner Chilcott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-02306
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Contraception
Keywords: Contraception
MeSH Terms: interventions — Norethindrone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Norethindrone 1 mg / ethinyl estradiol 20 mcg

SUMMARY:
This is an non-comparative study. There is no statistical hypothesis. The effects of extension of treatment on bleeding will be recorded and described.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 25-40
* History of regular cycles

Exclusion Criteria:

* Current or recent (within 2 months) users of hormonal contraceptives
* Contraindications for use of hormonal contraception
* Conditions which affect the absorption or metabolism of steroid hormones
* BMI > 35

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Number of bleeding/spotting days/episodes per treatment cycle

SECONDARY OUTCOMES:
Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Sponsor GmbH
Locations (21):
- United States (21):
  - Warner Chilcott Investigational Site, Phoenix, Arizona
  - Warner Chilcott Investigational Site, Tempe, Arizona
  - Warner Chilcott Investigational Site, Carmichael, California
  - Warner Chilcott Investigational Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Site, Leesburg, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, West Palm Beach, Florida
  - Warner Chilcott Investigational Site, Decatur, Georgia
  - Warner Chilcott Investigational Site, Roswell, Georgia
  - Warner Chilcott Investigational Site, Peoria, Illinois
  - Warner Chilcott Investigational Site, Lexington, Kentucky
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, New Bern, North Carolina
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Site, Greenville, South Carolina
  - Warner Chilcott Investigational Site, Pleasant Grove, Utah
  - Warner Chilcott Investigational Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Site, Sandy City, Utah
  - Warner Chilcott Investigational Site, Virginia Beach, Virginia
  - Warner Chilcott Investigational Site, Seattle, Washington